CLINICAL TRIAL: NCT01731964
Title: Pilot Study of WA-NG Telescope Prosthesis in Patients With Central Vision Impairment Associated With End-stage Age-related Macular Degeneration
Brief Title: Study of WA-NG Telescope Prosthesis in Patients With End-stage Age-related Macular Degeneration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA-NG-001 ASSAF HAROFEH
Record Dates: First submitted 2012-11-14; First posted 2012-11-22 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-04

CONDITIONS: Age Related Macular Degeneration
Keywords: Macular Degeneration; Visual Impairment; Implantable Telescope
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WA- NG Telescope Prothesis (Experimental): Implantable Miniature Telescope for end stage AMD
  Interventions: Device: Telescope prosthesis; Device: WA-NG Telescope Prothesis

INTERVENTIONS:
Device: Telescope prosthesis — Monocular implantation of the telescope prosthesis after cataract extraction
  Other Names: IMT-NG
Device: WA-NG Telescope Prothesis — The WA-NG telescope prosthesis (Figure 1) is the next generation telescopic implantable device which, when combined with the optics of the cornea, constitutes a telephoto system for improvement of visual acuity in patients with severe to profound vision impairment due to bilateral, end-stage age-related macular degeneration. The device is implanted in one of the patient's eyes. In this way, the implanted eye provides central vision and the non-implanted eye can continue to provide peripheral vision.

SUMMARY:
This is a pilot study to evaluate the safety of the Model WA-NG telescope prosthesis in patients with bilateral moderate to profound central vision impairment due to end-stage age-related macular degeneration.

DETAILED DESCRIPTION:
Patients will be screened for eligibility and informed consent will be obtained from those who meet screening criteria and are interested in participating in the study. Eligible patients will be examined preoperatively to obtain a medical history and to establish a baseline for ocular condition. Baseline measurements will include successful use of an external telescope.

Postoperatively, patients will undergo ophthalmic evaluation at regular intervals as specified in this protocol and will be required to return for 6 to 10 additional visits for vision training with a low vision specialist.

ELIGIBILITY:
Inclusion Criteria:

Bi-lateral, stable, moderate to profound (20/80 to 20/800) central vision impairment due to bilateral scotoma associated with end-stage macular degeneration, defined as retinal finds of bilateral, geographic atrophy or disciform scar with foveal involvment. Phakic in the operative eye. Must achieve a 5 letter improved with external telescope simulator.

Exclusion Criteria:

Evidence of active CNV or any ophthalmic pathology that compromises peripheral vision of fellow eye or predisposes eye rubbing. Previous intraocular of corneal surgery of any kind in operative eye. Retinal disease, optic nerve disease, diabetic retinopathy, retinal tears, or any introcular tumor or medical or ophthalmic condition that in the opinion of the investigator renders the subject unsuitable for participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 12 months
  Positional stability assessed by slit lamp examination and anterior segment OCT

SECONDARY OUTCOMES:
Safety | 12 months
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Avni, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel